CLINICAL TRIAL: NCT04184245
Title: Cardiovascular and Cerebrovascular Responses to Cardio-respiratory Events in Very Preterm Infants During the Transitional Period
Brief Title: Hemodynamic Responses to Cardio-respiratory Events in Preterm Infants
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Luigi Corvaglia, Associate Professor, Neonatal Consultant, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: SO-CRE-2
Record Dates: First submitted 2019-11-29; First posted 2019-12-03 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Apnea of Prematurity; Preterm Birth; Patent Ductus Arteriosus; Hypoxia, Brain; Cardiac Output, Low; Bradycardia Neonatal; Hypoxia Neonatal
Keywords: preterm infants; hypoxic episodes; non-invasive cardiac output monitoring; near infrared spectroscopy; cardiac output; cerebral oxygenation; bradycardia; cardiorespiratory events
MeSH Terms: conditions — Apnea; Premature Birth; Ductus Arteriosus, Patent; Hypoxia, Brain; Cardiac Output, Low; Asphyxia Neonatorum; Bradycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Intermittent episodes of hypoxemia and/or bradycardia, also defined as cardio-respiratory events (CRE) are very frequent in preterm infants and may result in transient hypoxia and hypoperfusion of target organs, with possible clinical implications. The hemodynamic instability that characterizes the first 72 hours of life, also called as transitional period, place preterm infants at high risk of complications and may contribute to enhance fluctuations in end-organ perfusion and oxygenation induced by CRE. In this study we aimed to explore cardiovascular and cerebrovascular changes determined by different CRE types in preterm infants during the transitional period.

DETAILED DESCRIPTION:
Intermittent episodes of hypoxemia and/or bradycardia, also defined as cardio-respiratory events (CRE) are very frequent in preterm infants and may result in transient hypoxia and hypoperfusion of target organs, with possible clinical implications. The hemodynamic instability that characterizes the first 72 hours of life, also called as transitional period, place preterm infants at high risk of complications and may contribute to enhance fluctuations in end-organ perfusion and oxygenation induced by CRE. Moreover, during this period, several clinical variables (e.g., antenatal steroid administration, gestational age [GA], patent ductus arteriosus [PDA], respiratory support etc.) may contribute to modulate the hemodynamic fluctuations in response to CRE.

Hence, this study aims:

* to explore changes in the main cardiovascular and cerebrovascular parameters elicited by different CRE types
* to evaluate whether different antenatal, perinatal and postnatal factors may influence the observed cardiovascular and cerebrovascular responses to CRE.

Infants born at S. Orsola-Malpighi Hospital are consecutively enrolled in this observational, prospective study if fulfilling the following eligibility criteria: gestational age (GA) <32 weeks' gestation, birth weight <1500 g, 0-12 hours of life, written informed consent obtained from the parents/legal guardians of each infant.

As routinely performed in infants with the eligible characteristics, the enrolled infants undergo a simultaneous, continuous and non-invasive monitoring of

* peripheral oxygen saturation (SpO2) and heart rate (HR) using a pulse oximeter
* cerebral tissue oxygenation index (cTOI) and cerebral total hemoglobin index (cTHI), which represents a proxy of cerebral blood flow, using near infrared spectroscopy. Cerebral fraction of oxygen extraction (cFTOE) is also calculated as follows: (SpO2-cTOI)/SpO2.
* cardiovascular parameters (cardiac output [CO], stroke volume [SV], cardiac contractility index [ICON], systemic vascular resistance [SVR]) using electrical cardiometry.

In the enrolled infants, each monitoring device is connected via a RS232 cable to a laptop running ICM+® (https://icmplus.neurosurg.cam.ac.uk/, Cambridge Enterprise, UK), a software tool that allows a real-time synchronized multi-parametric data collection, which recorded the above mentioned parameters continuously, from the time of enrollment up to 72 hours of life.

Cardiorespiratory event types are classified on the basis of SpO2 and HR values as follows:

* isolated desaturation (ID): SpO2 <85% and classified into mild (SpO2 80-84%), moderate (SpO2 70-79%) and severe (SpO2 <70%).
* isolated bradycardia (IB): any HR drop <100 bpm or >30% from baseline values, calculated daily over the first 72 hours of life
* desaturation and bradycardia occurring within a 60-sec time window: combined events (DB).

The following antenatal and neonatal data are tracked down on a specific case report form: GA, antenatal steroids (complete course vs. incomplete course or not given) evidence of reversed end-diastolic flow at antenatal umbilical Doppler (uREDF) (present vs. absent); ventilatory status over the first 72 hours of life (continuous positive airway pressure [CPAP] vs. nasal cannulas or self-ventilating in air [SVIA]); surfactant administration; development of IVH over the first 72 hours of life.

A screening echocardiogram is routinely performed at the time of enrollment and repeated 6-12 hourly in the presence of a patent ductus arteriosus (PDA) or 12-24 hourly if there is no evidence of PDA. Based on echocardiographic features, the ductal status is classified as follows: no evidence of PDA (noPDA), restrictive PDA (rPDA; restrictive shunt pattern and left atrium to aortic root ratio [LA:Ao] ratio <1.5), hemodynamically significant PDA (hsPDA; pulsatile shunt pattern, LA:Ao ratio ≥1.5 or presence of reversed end-diastolic flow either in the descending aorta or in the anterior cerebral artery).

For statistical analysis, percentage changes of cardiovascular (CO, ICON, SVR) and cerebrovascular (cTOI, cTHI, cFTOE) parameters will be compared between different CRE types (ID, DB and IB) using Kruskal-Wallis test. Generalized estimating equation (GEE) models will be used to analyze the concomitant effect of clinical variables (e.g., GA, uREDF, antenatal steroids, ductal and ventilatory status etc.) on the percentage changes of the study parameters. IBM SPSS, version 25.0, will be used for statistical analysis. The significance level is set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* gestational age <32 weeks' gestation AND/OR birth weight <1500 g

Exclusion Criteria:

* major congenital malformations
* congenital heart disease
* mechanical ventilation

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants on spontaneous breathing during the transitional period (0-72 hours of life).
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-03 (Actual)

PRIMARY OUTCOMES:
Increase/reduction of cTOI during isolated desaturation, isolated bradycardia and desaturation-bradycardia | 0-72 hours of life
  Comparison of percentage cTOI changes (cTOI at baseline/during the event) among isolated desaturation, isolated bradycardia and desaturation-bradycardia
Increase/reduction of cFTOE during isolated desaturation, isolated bradycardia and desaturation-bradycardia | 0-72 hours of life
  Comparison of percentage cFTOE changes (baseline/during the event) among isolated desaturation, isolated bradycardia and desaturation-bradycardia
Increase/reduction of cTHI during isolated desaturation, isolated bradycardia and desaturation-bradycardia | 0-72 hours of life
  Comparison of percentage cTHI changes (baseline/during the event) among isolated desaturation, isolated bradycardia and desaturation-bradycardia
Increase/reduction of CO during isolated desaturation, isolated bradycardia and desaturation-bradycardia | 0-72 hours of life72 hours
  Comparison of percentage CO changes (CO at baseline/during the event) among isolated desaturation, isolated bradycardia and desaturation-bradycardia
Increase/reduction of SV during isolated desaturation, isolated bradycardia and desaturation-bradycardia | 0-72 hours of life
  Comparison of percentage SV changes (baseline/during the event) among isolated desaturation, isolated bradycardia and desaturation-bradycardia
Increase/reduction of ICON during isolated desaturation, isolated bradycardia and desaturation-bradycardia | 0-72 hours of life
  Comparison of percentage ICON changes (baseline/during the event) among isolated desaturation, isolated bradycardia and desaturation-bradycardia
Increase/reduction of SVR during isolated desaturation, isolated bradycardia and desaturation-bradycardia | 0-72 hours of life
  Comparison of percentage SVR changes (baseline/during the event) among isolated desaturation, isolated bradycardia and desaturation-bradycardia

SECONDARY OUTCOMES:
Effect of neonatal characteristics on cerebrovascular parameters | 0-72 hours of life
  Generalized estimating equation (GEE) analysis evaluating the effect of clinical variables (e.g., GA, uREDF, antenatal steroids, ductal and ventilatory status etc.) on percentage changes of cTOI, cFTOE, cTHI.
Effect of neonatal characteristics on cardiovascular parameters | 0-72 hours of life
  Generalized estimating equation (GEE) analysis evaluating the effect of clinical variables (e.g., GA, uREDF, antenatal steroids, ductal and ventilatory status etc.) on percentage changes of CO, SV, ICON, SVR

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Corvaglia, MD, Principal Investigator — S. Orsola-Malpighi University Hospital, Bologna, Italy
Locations (1):
- S. Orsola-Malpighi University Hospital, Bologna, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: No